CLINICAL TRIAL: NCT00065052
Title: Modifying the Home Television Watching Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MODHTV (completed); 1R01DK063442 (NIH)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Body Weight Changes
Keywords: physical activity; television; child obesity; Reduce TV; Usual control
MeSH Terms: conditions — Obesity; Body Weight Changes; Motor Activity; Pediatric Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior modification

SUMMARY:
The purpose of this study is to determine if limiting television (TV) and computer time will result in a stabilization or smaller increase in body mass index (BMI), lower energy intake, and increased physical activity in 4-7 year old obese (>85th BMI percentile) children over two years.

DETAILED DESCRIPTION:
There is a positive correlation between obesity and television watching in adults and children. And, television watching, controlling for current obesity, is a predictor of future obesity. Almost half of all children watch 3 or more hours of television each day. The American Academy of Pediatrics recommends that children watch no more than 1-2 hours each day.

Families will be randomized to one of two conditions. Half the families will be taught to use the TV Allowance to reduce their child's TV and computer use by one-half over a six month period and the other half will use the device to monitor TV watching (control group). This study uses TV Allowance units to monitor home television watching, video game playing, and computer use. The TV Allowance can also be used to limit the amount of TV and computer use by programming it to allow a specific number of hours for each family member. Heights, weights, food intake, and physical activity will be measured at baseline and every six months. The purpose of this study is to determine if limiting television and computer time will result in a stabilization or smaller increase in BMI, lower energy intake, and increased physical activity in 4-7 year old obese (>85th BMI percentile) children over two years.

ELIGIBILITY:
* Greater than the 85th BMI percentile
* Minimum of 15 hours of TV watching, computer use, and video game playing per week
* No medical conditions that may affect the child's ability to safely participate in physical activity

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2002-09; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H. Epstein, Ph.D., Principal Investigator — State Universtiy of New York at Buffalo, Department of Pediatrics
Locations (1):
- University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Epstein LH, Roemmich JN, Robinson JL, Paluch RA, Winiewicz DD, Fuerch JH, Robinson TN. A randomized trial of the effects of reducing television viewing and computer use on body mass index in young children. Arch Pediatr Adolesc Med. 2008 Mar;162(3):239-45. doi: 10.1001/archpediatrics.2007.45. PMID 18316661